CLINICAL TRIAL: NCT02559726
Title: Identification and Quantification of a Mechanical Hyper-synchronicity State in Hypertrophic Cardiomyopathy (HCM) With Left Outflow-tract Obstruction and Description of Its Electrical and Electro-mechanical Characteristics Thanks to an Innovative Multi-imaging Approach to Predict a Positive Response to Dual Chamber Pacing. The Hsync Study.
Brief Title: Hyper-synchronicity in Hypertrophic Cardiomyopathy (HCM) : Description, Mechanism and Origin With a Multi-imaging Approach to Predict Dual Chamber Pacing Response
Acronym: HSYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2014/06
Record Dates: First submitted 2015-06-26; First posted 2015-09-24 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Hypertrophic Cardiomyopathy; Mechanical Hyper-synchronicity
Keywords: Hypertrophic cardiomyopathy, hyper-synchronicity, outflow-tract obstruction, dual chamber pacing
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- O-HCM (Experimental): 20 patients with Hypertrophic Cardiomyopathy with outflow-tract obstruction
  Interventions: Procedure: Echocardiography (TEE); Device: Magnetic resonance imaging (MRI) with gadolinium enhancement; Procedure: 3D electrocardiographic mapping (ECM)
- NO-HCM (Experimental): 20 patients with Hypertrophic Cardiomyopathy without outflow-tract obstruction
  Interventions: Procedure: Echocardiography (TEE); Device: Magnetic resonance imaging (MRI) with gadolinium enhancement; Procedure: 3D electrocardiographic mapping (ECM)
- healthy volunteers (Other): 20 healthy volunteers
  Interventions: Procedure: Echocardiography (TEE); Device: Magnetic resonance imaging (MRI) without gadolinium enhancement; Procedure: 3D electrocardiographic mapping (ECM)

INTERVENTIONS:
Procedure: Echocardiography (TEE)
Device: Magnetic resonance imaging (MRI) with gadolinium enhancement
  Arms: NO-HCM; O-HCM
Device: Magnetic resonance imaging (MRI) without gadolinium enhancement
  Arms: healthy volunteers
Procedure: 3D electrocardiographic mapping (ECM)
  Other Names: 3-dimensional electrocardiographic mapping (ECM) combined with computed tomography-scan

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a common genetic cardiovascular disease. Outflow-tract gradient of 30 mmHg or more under resting conditions is an independent determinant of symptoms of progressive heart failure and death.

The investigators hypothesize that the electrical approach by dual chamber pacing could improve symptoms and reduce outflow-tract obstruction in a specific sub-group of selected patients with a mechanical hyper-synchronicity. The aim of the study is to identify and describe this phenomenon in HCM with (O-HCM) and without (NO-HCM) outflow-tract obstruction thanks to innovative multi-imaging approach.

DETAILED DESCRIPTION:
The concept of physiological ventricular desynchrony was described recently with technics of myocardial deformation analysis applied in animal models. Authors confirmed the existence of a time delay in the contraction of the apical walls before basal walls. In O-HCM, the outflow-tract obstruction could be explained by a mechanical hyper-synchronicity between apical and basal walls. This study aims to describe the possible hyper-synchronized contraction in O-HCM and NO-HCM patients unlike the physiological desynchrony observed in healthy volunteers (HV) For this purpose, three imaging tests will be used at baseline: echocardiography (TEE), magnetic resonance imaging (MRI) with gadolinium enhancement only in HCM, and 3-dimensional electrocardiographic mapping (ECM) combined with computed tomography-scan. No follow-up is planned for this study.

ELIGIBILITY:
Inclusion Criteria:

* HCM: Adults aged more than 18 years with sarcomeric hypertrophic cardiomyopathy under optimal medical therapy, isolated septal hypertrophy, sinus rhythm, exploitable acoustic window. For women of childbearing age, effective contraception and required negative pregnancy test.
* O-HCM : outflow-tract gradient more than 30 mmHg at rest and during exercise
* NO-HCM : outflow-tract gradient less than 30 mmHg at rest and during exercise
* HV: Adults aged more than 18 years, without cardiovascular disease. For women of childbearing age, effective contraception and required negative pregnancy test.

Exclusion Criteria:

- HV: unusable acoustic window

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
Mechanical time delay in contraction between basal and apical walls in TEE and MRI in O-HCM, NO-HCM and healthy volunteers | Day 1
  The main interest variable is the delay value (ms) of the contraction between basal and apical walls measured by TEE and MRI.

SECONDARY OUTCOMES:
Relationship between each mesure with hyper-synchronicity and outflow-tract gradient | Day 1
Electrical time delay in ECM between basal and apical walls and relationship with hyper-synchronicity and outflow tract gradient. | Day 1
Mechanical time delay between septal and lateral walls in MRI and TEE. | Day 1
Evolution of mechanical time delay between basal and apical walls at rest and exercise in O-HCM and NO-HCM and relationship with outflow-tract gradient. | Day 1
Delay between peaks of basal and apical radial displacement in MRI | Day 1
Delay between the beginning of the apical and basal radial displacement in MRI | Day 1
Apical-basal phase on a phase analysis of the radial displacement data in MRI | Day 1
Delay between apical and basal peaks circumferential strain in MRI | Day 1
Delay between the beginning of the apical and basal circumferential deformation in MRI | Day 1
Twist angle between the base and the apex in MRI | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Claire CORNOLLE, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Reant P, Bonnet G, Dube F, Massie C, Reynaud A, Michaud M, Duchateau J, Lafitte S. Hypersynchrony in sarcomeric hypertrophic cardiomyopathy: description and mechanistic approach using multimodal electro-mechanical non-invasive cartography (HSYNC study). Front Cardiovasc Med. 2024 Jun 7;11:1359657. doi: 10.3389/fcvm.2024.1359657. eCollection 2024. PMID 38911519